CLINICAL TRIAL: NCT04627558
Title: Validity Reliability of The Dubousset Functional Test in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Yusuf Emre Bozkurt, Principal Investigator, Kırıkkale University
Other Study IDs: Dubousset Functional Test
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Stroke Syndrome; Balance; Distorted; Walking, Difficulty
MeSH Terms: conditions — Stroke; Mobility Limitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke patients, balance assessment: Dubousset Function Test, 3-m backwards walk test, timed up and go test,Tinnetti Balance and Gait Test, Berg BalanceTest, Functional Reach Test
  Interventions: Other: stroke patients, balance assessment

INTERVENTIONS:
Other: stroke patients, balance assessment — validity relability dubousset functional test

SUMMARY:
Increased muscle tone, decreased normal range of motion, and functional impairments may result in decreased load on the affected limb, deviations in gait patterns, balance and coordination disorders in individuals with stroke.

In the literature, there are many scales that evaluate balance and functional performance in stroke. However there is no validity and reliability study of Dubousset Function Test developed to evaluate balance and functional performance of stroke. For this reason, the aim of study is to examine the validity and reliability of Dubousset Function Test in stroke patients.

DETAILED DESCRIPTION:
While the ambulation ability is completely lost in some patients after stroke, impaired balance reactions and increased postural oscillations cause an increase in the fear of falling and the risk of falling in stroke patients. These disturbances cause stroke patients to make more effort to balance while standing. Balance assessment performed in individuals with stroke determines the risk of falling and is important in preventing complications that may develop due to loss of balance.

Dubousset Functional Test (DFT); A conceptually practical four-component assessment test has been proposed by Dr. Jean Dubousset to assess the functional capacity of adult individuals. The validity of the test was made in individuals with spinal deformity. DFT; It consists of four components: getting up from a chair without arms and walking 5 meters forward and backward, descending and climbing steps, transition from standing to sitting on the ground, and the dual task test in which the individual walks while counting down from 50 at the same time. In the literature, there are many scales that evaluate balance and functional performance in stroke. However there is no validity and reliability study of Dubousset Function Test developed to evaluate balance and functional performance of stroke. For this reason, the aim of study is to examine the validity and reliability of Dubousset Function Test in stroke patients

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,

  * Getting a diagnosis of stroke,
  * Not having cooperation and communication problems
  * To be able to walk 10 m independently with or without device

Exclusion Criteria:

* Have a neurological or orthopedic problem other than stroke that will affect functionality and balance
* Individuals with contraindications for advanced cardiovascular disease and mobilization will not be included in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Dubousset Function Test | First day
  The four components of the DFT included (1) the Up Walking Test: participants rose without assistance from a and seated position in a chair that did not have arms, walked 5 meters (500 cm) forward before stopping, walked backwards 5 meters, and sat again without assistance; (2) the Steps Test: from a starting position 50 cm away, volunteers climbed three stairs, turned around on the third step (top), and walked down the three steps; (3) Down and Sitting Test: from a standing position, participants sat on the ground and stood up again, using assistance as needed; (4) Dual-Tasking Test: participants walked 5 meters forward, turned around, and walked 5 meters back to the starting position while performing a working memory test (counting down from 50 by intervals of 2).
timed up and go test | first day
  A standard chair is used for testing. First, the patient is asked to sit on the chair. The patient is then asked to stand up and walk regularly at a distance of 3 meters with a predetermined length, then return to the chair after 3 meters
3-m backwards walk test | first day
  A distance of 3 m is measured and marked with black tape. Individuals are asked to follow the heel and black band.
  With the 'start' command they are asked to walk backwards quickly. When the distance of 3 m is completed, a stop is instructed. Individuals are not allowed to run during the test. They are allowed to look back if they wish. The assessor walks behind individuals throughout the test. The test is repeated 3 times, the averages are recorded
Tinetti Balance and Gait Test | first day
  In the test used to evaluate balance, walking score is maximum 12 points, balance score is maximum 16 points and a total of 28 points.
Berg Balance Test | first day
  The BBS consists of 14 items to directly monitor the maintenance of body balance during performance
Funtional Reach Test | first day
  It is used to measure both the balance of the individual functionally and the amount of dynamic reach

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Emre Bozkurt, PT, Principal Investigator — Kırıkkale University
Locations (1):
- Yusuf Emre Bozkurt, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diebo BG, Challier V, Shah NV, Kim D, Murray DP, Kelly JJ, Lafage R, Paulino CB, Passias PG, Schwab FJ, Lafage V. The Dubousset Functional Test is a Novel Assessment of Physical Function and Balance. Clin Orthop Relat Res. 2019 Oct;477(10):2307-2315. doi: 10.1097/CORR.0000000000000820. PMID 31135543